CLINICAL TRIAL: NCT03549429
Title: A Randomized Control Trial of Tegaderm vs. EyeGard for Eye Protection During General Anesthesia
Brief Title: Tegaderm vs. EyeGard for Eye Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12884
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Intervention Model Description: Every patient will have each tape on each eye -EyeGard® on one eye and the TegadermTM on the other eye according to the randomization schema.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TegadermTM on R eye, EyeGard® on L eye (Experimental): Patients will get TegadermTM on Right eye, EyeGard® on Left eye
  Interventions: Device: Medical tapes: TegadermTM and EyeGard®
- TegadermTM on L eye, EyeGard® on R eye (Experimental): Patients will get TegadermTM on Left eye, EyeGard® on Right eye
  Interventions: Device: Medical tapes: TegadermTM and EyeGard®

INTERVENTIONS:
Device: Medical tapes: TegadermTM and EyeGard® — TegadermTM and EyeGard® will be placed over patients' eyes during surgery with general anesthesia.

SUMMARY:
This study compares TegadermTM and EyeGard® in general anesthesia.

DETAILED DESCRIPTION:
Protective eye tape is used during anesthesia in order to prevent corneal abrasion and other eye injuries. However, there is no single accepted practice of how to protect the eyes during anesthesia, and a variety of different tapes and techniques have been adopted in different institutions. In this study, investigators will compare two tapes, TegadermTM and EyeGard® to determine if one is less likely to cause eyelid irritation in an effort to improve care for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Surgeries scheduled for anesthesia of any duration

Exclusion Criteria:

* Any patient that does not consent
* Any patient who has:
* Pre-existing eyelid erythema or other eyelid trauma
* Eyelid piercings
* Any surgery on the head, brain, neck, teeth, mouth, eyes or face
* Surgery in the prone position
* Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Drzymalski, MD, Principal Investigator — Tufts Medical Center Dept. of Anesthesia
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Drzymalski DM, Ward K, Hernandez JM, Hoot J, Au SC, Yang FC, Azocar RJ. The effect of Tegaderm versus EyeGard(R) on eyelid erythema during general anesthesia: a randomized-controlled trial. Can J Anaesth. 2020 May;67(5):560-567. doi: 10.1007/s12630-020-01588-6. Epub 2020 Feb 13. PMID 32095992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 159 patients were enrolled (consented) but not randomized. The reasons for not randomizing include:
  * Research assistant unavailable (n=6)
  * Anesthetic plan change (n=4)
  * Surgical plan change (n=4)
  * Tape sensitivity (n=1)
Period: Overall Study
Arm/Group | TegadermTM on R Eye, EyeGard® on L Eye | TegadermTM on L Eye, EyeGard® on R Eye
Started | 81 | 78
Completed | 76 | 75
Not Completed | 5 | 3
Not completed — Protocol Violation | 5 | 3

BASELINE CHARACTERISTICS:
Population: Those who were eligible were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | TegadermTM on R Eye, EyeGard® on L Eye | TegadermTM on L Eye, EyeGard® on R Eye | Total
Number analyzed (Participants) | 81 | 78 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 29 | 50
  >=65 years | 60 | 49 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 40 | 33 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 40 | 33 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 65 | 60 | 125
  Non-Caucasian | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Eyelid Erythema
Description: The amount of erythema caused upon removal of the tape is the primary outcome of interest. Investigators will use the following 0-3 tape-associated skin index grading scale to grade eyelid erythema:
  0- no erythema
  1. mild erythema
  2. moderate erythema
  3. severe erythema The primary outcome will then be converted to a binary scale (0= no erythema, 1= erythema) for the purposes of analysis.
Time Frame: Standardized photos will be taken within 5 minutes of removing tape after surgery (surgery of any duration)
Population: Inclusion Criteria: Age ≥ 18, surgeries scheduled for anesthesia of any duration.
  Exclusion Criteria: Any patient that does not consent, any patient who has pre-existing eyelid erythema or other eyelid trauma/piercings, any surgery on the head, brain, neck, teeth, mouth, eyes or face, surgery in the prone position, patients <18 years old
Measure: Count of Participants; unit: Participants
Groups:
- Erythema With TegadermTM Only; Erythema With EyeGard® Only: TegadermTM and EyeGard® will be placed over patients' eyes during surgery with general anesthesia. Half of the participants (n=76) will receive TegadermTM over their right eyelid and EyeGard over the left eyelid. The other half of the participants (n=75) will receive TegadermTM over their left eyelid and EyeGard over the right eyelid.
Arm/Group | Erythema With TegadermTM Only | Erythema With EyeGard® Only
Number analyzed (Participants) | 151 | 151
Participants | 117 | 105
Statistical Analysis 1: Comparison: Erythema With TegadermTM Only vs Erythema With EyeGard® Only; We compared the proportion of patients who had postoperative eyelid erythema with Tegaderm™ to those who had postop eyelid erythema with EyeGard®; Test type: Superiority; p = 0.03, McNemar; Percent difference = 8.0, 95% CI 2-sided [1.5 to 14.4]

2. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction will be based on one question and graded on a Likert Scale from 1-5. A score of 5 is considered better (higher satisfaction), while a 1 is considered lower. There are no subscales.
Time Frame: post-operation
Measure: Mean (Standard Deviation); unit: Units on a scale of 1-5
Groups:
- TegadermTM: TegadermTM and EyeGard® will be placed over patients' eyes during surgery with general anesthesia. Half of the participants (n=76) will receive TegadermTM over their right eyelid and EyeGard over the left eyelid. The other half of the participants (n=75) will receive TegadermTM over their left eyelid and EyeGard over the right eyelid.
- EyeGard®: TegadermTM and EyeGard® will be placed over patients' eyes during surgery with general anesthesia. TegadermTM and EyeGard® will be placed over patients' eyes during surgery with general anesthesia. Half of the participants (n=76) will receive TegadermTM over their right eyelid and EyeGard over the left eyelid. The other half of the participants (n=75) will receive TegadermTM over their left eyelid and EyeGard over the right eyelid.
Arm/Group | TegadermTM | EyeGard®
Number analyzed (Participants) | 151 | 151
Units on a scale of 1-5 | 4.94 (0.42) | 4.91 (0.51)
Statistical Analysis 1: Comparison: TegadermTM vs EyeGard®; Test type: Superiority; p = 0.23, t-test, 2 sided; paired; Mean Difference (Final Values) = 0.03

3. Secondary Outcome: Rate of Corneal Abrasions
Description: Corneal abrasion is assessed in the recovery room
Time Frame: post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | TegadermTM | EyeGard®
Number analyzed (Participants) | 151 | 151
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: For the length of participation in the study; approx. 3-10 hours
Description: This study does not pose any additional safety risks beyond those associated with the application of protective tape over the patient's eyelids that occurs during standard surgical procedures. These risks include injury to the eyelid such as mild to severe erythema, edema, and abrasion.
Arm/Group | TegadermTM on R Eye, EyeGard® on L Eye | TegadermTM on L Eye, EyeGard® on R Eye
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/159
Other Adverse Events (participants affected / at risk) | 0/159 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03549429/Prot_SAP_001.pdf